CLINICAL TRIAL: NCT03233529
Title: A PHASE 2A, RANDOMIZED, DOUBLE-BLIND, VEHICLE-CONTROLLED STUDY, TO CHARACTERIZE THE MECHANISM OF ACTION OF CRISABOROLE OINTMENT 2%, BY EVALUATION OF EFFICACY AND CHANGES IN SKIN BIOMARKERS, IN ADULT SUBJECTS WITH MILD TO MODERATE ATOPIC DERMATITIS, WITH A 4 WEEK OPEN-LABEL EXTENSION
Brief Title: Crisaborole Ointment 2% Skin Biomarker Biopsy Study in Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: C3291001
Record Dates: First submitted 2017-07-12; First posted 2017-07-28 (Actual); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis; atopic eczema; eczema; topical treatment; skin diseases; phosphodiesterase-4 inhibitor; PDE-4 inhibitor; crisaborole
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Skin Diseases | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Crisaborole ointment (Experimental)
  Interventions: Drug: Crisaborole ointment 2% BID
- Placebo ointment (vehicle) (Placebo Comparator)
  Interventions: Drug: Placebo ointment (vehicle)

INTERVENTIONS:
Drug: Crisaborole ointment 2% BID — Crisaborole ointment 2% BID for 15 days (double blind); additional 28 days (open label)
  Arms: Crisaborole ointment
Drug: Placebo ointment (vehicle) — Placebo ointment (vehicle) BID for 15 days (double blind)
  Arms: Placebo ointment (vehicle)

SUMMARY:
This study is being conducted to characterize the mechanism of action of crisaborole ointment 2%, by evaluation of efficacy and changes in key skin biomarkers in atopic dermatitis (AD) lesions treated with crisaborole ointment 2% over vehicle, in subjects with mild to moderate AD. Two identified AD skin lesions for each subject will be treated for the first 15 days, one with crisaborole ointment 2% and one with vehicle, in a blinded manner, and biopsies for biomarker analysis will be performed on the lesions. Following completion of the blinded treatment period, subjects will start the 28 day open label period during which all AD affected skin lesions will be treated with crisaborole ointment 2% twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of active atopic dermatitis (AD) with at least 6 month history prior to Screening and that has been clinically stable for 1 month.
* Investigator's Static Global Assessment (ISGA) of 2 (mild) or 3 (moderate) at Baseline.
* Body surface area (BSA) covered with AD of at least 0.5% and no more than 10% at Baseline, calculation excluding face, scalp, axilla, genitals, groin area, palms, back of the hands, and soles.
* Two lesions of AD at least 3 cm x 3 cm in size and at least 5 cm apart, with identical Lesion ISGA score of greater than/equal to 3.

Exclusion Criteria:

* Clinically infected AD or requires high potency topical corticosteroids or systemic (oral/injectable) corticosteroids to manage AD.
* History of angioedema or anaphylaxis to topical products or known sensitivity to components of crisaborole ointment 2%.
* History of cancer (except squamous or basal cell carcinoma or carcinoma in situ of the skin).
* Previous treatment with any topical or systemic PDE4 inhibitor unless stopped for the reason of lack of efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Innovaderm Research Incorporated, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Bissonnette R, Pavel AB, Diaz A, Werth JL, Zang C, Vranic I, Purohit VS, Zielinski MA, Vlahos B, Estrada YD, Saint-Cyr Proulx E, Ports WC, Guttman-Yassky E. Crisaborole and atopic dermatitis skin biomarkers: An intrapatient randomized trial. J Allergy Clin Immunol. 2019 Nov;144(5):1274-1289. doi: 10.1016/j.jaci.2019.06.047. Epub 2019 Aug 13. PMID 31419544
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C3291001&StudyName=A+Phase+2%2C+Single-center%2C+Randomized%2C+Double-blind+Study+To+Explore+The+Mechanism+Of+Action+Of+Crisaborole+Topical+Ointment+2%25+In+Patients+With+Atopic+Dermatitis
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C3291001&StudyName=A+Phase+2a%2C+Randomized%2C+Double-blind%2C+Vehicle-controlled+Study%2C+To+Characterize+The+Mechanism+Of+Action+Of+Crisaborole+Ointment+2%25%2C+By+Evaluation+Of+Efficacy+And+Changes+In+Skin+Biomarkers%2C+In+Adult+Subjects+With+Mild+To+Moderate+Atopic+Dermatitis%2C+With+A+4+Week+Open-label+Extension

RESULTS

PARTICIPANT FLOW:
Groups:
- Crisaborole Ointment 2%+Vehicle, Then Crisaborole Ointment 2%: The study consisted of 2 periods, i.e., a double-blind period from Day 1 to Day 15 skin biopsy collection, and an open-label period from Day 15 skin biopsy collection to the end of study (Day 71). Each participant received double-blind topical administration of crisaborole ointment 2 percent (%) for 1 target lesion and placebo ointment vehicle (referred to as vehicle) for the other target lesion (i.e., each participant was treated with both crisaborole and vehicle), twice daily from Day 1 to Day 14; then received open-label topical administration of crisaborole ointment 2% for all atopic dermatitis skin areas (excluding scalp) twice daily from Day 15 to Day 42.
Period: Double-Blind Period (Day 1 to Day 15)
Arm/Group | Crisaborole Ointment 2%+Vehicle, Then Crisaborole Ointment 2%
Started | 40
Completed | 39
Not Completed | 1
Not completed — Adverse Event | 1
Period: Open-Label Period (Day 15 to Day 71)
Arm/Group | Crisaborole Ointment 2%+Vehicle, Then Crisaborole Ointment 2%
Started | 39
Completed | 38
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of investigational product.
Arm/Group | Crisaborole Ointment 2%+Vehicle, Then Crisaborole Ointment 2%
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lesion Total Sign Score (TSS) for Target Lesions Treated With Crisaborole Ointment 2% or Vehicle at Day 15
Description: The lesion TSS is an assessment of target lesion severity based on the severity of the following 4 clinical signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification, each of which was rated on a scale of 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe). These 4 ratings were then added to create the TSS, which ranges from 0 (none) to 12 (most severe), with higher score representing greater severity.
Time Frame: Baseline (Day 1), Day 15
Population: All randomized participants who received at least 1 dose of investigational product and had TSS assessment at Day 15.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Crisaborole Ointment 2% Treated Lesion: On Days 1 to 14, for each participant, one target lesion was treated with crisaborole ointment 2% and the other target lesion was treated with vehicle, i.e., each participant was treated with both crisaborole and vehicle. This reporting group represents the target lesions that were treated with crisaborole ointment 2% during Days 1 to 14.
- Vehicle Treated Lesion: On Days 1 to 14, for each participant, one target lesion was treated with crisaborole ointment 2% and the other target lesion was treated with vehicle, i.e., each participant was treated with both crisaborole and vehicle. This reporting group represents the other target lesions that were treated with vehicle during Days 1 to 14.
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
units on a scale | -4.5 (0.31) | -2.1 (0.35)
Statistical Analysis 1: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -2.4, 95% CI 2-sided [-3.1 to -1.7], Standard Error of Mean 0.35

2. Primary Outcome: Change From Baseline in Key Skin Biomarker Chemokine Ligand (CCL)17 Expression in Target Lesions Treated With Crisaborole Ointment 2% or Vehicle at Day 15
Description: CCL17 is one of the key skin biomarkers of atopic dermatitis. Expression levels tested by Taqman low density array (TLDA) reverse-transcriptase (RT) polymerase chain reaction (PCR) were normalized to the housekeeping gene ribosomal protein lateral stalk subunit P0 (RPLP0) and log2-transformed prior to analysis.
Time Frame: Baseline (Day 1), Day 15
Population: All randomized participants who received at least 1 dose of investigational product, with both Day 1 and Day 15 biopsies done, and without protocol violations that were thought to impact the biomarker expression during the double-blind vehicle-controlled period.
Measure: Mean (Standard Error); unit: log2(normalized expression)
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
log2(normalized expression) | -1.2787 (0.36339) | -0.2881 (0.34055)
Statistical Analysis 1: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p = 0.0420, Mixed Models Analysis; Least Squares Mean Difference = -0.9906, Standard Error of Mean 0.48404

3. Primary Outcome: Change From Baseline in Key Skin Biomarker CCL18 Expression in Target Lesions Treated With Crisaborole Ointment 2% or Vehicle at Day 15
Description: CCL18 is one of the key skin biomarkers of atopic dermatitis. Expression levels tested by TLDA RT PCR were normalized to the housekeeping gene RPLP0 and log2-transformed prior to analysis.
Time Frame: Baseline (Day 1), Day 15
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log2(normalized expression)
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
log2(normalized expression) | -0.7295 (0.25784) | -0.1849 (0.25272)
Statistical Analysis 1: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p = 0.1519, Mixed Models Analysis; Least Squares Mean Difference = -0.5446, Standard Error of Mean 0.37855

4. Primary Outcome: Change From Baseline in Key Skin Biomarker CCL22 Expression in Target Lesions Treated With Crisaborole Ointment 2% or Vehicle at Day 15
Description: CCL22 is one of the key skin biomarkers of atopic dermatitis. Expression levels tested by TLDA RT PCR were normalized to the housekeeping gene RPLP0 and log2-transformed prior to analysis.
Time Frame: Baseline (Day 1), Day 15
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log2(normalized expression)
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
log2(normalized expression) | -1.3267 (0.24359) | -0.1994 (0.22335)
Statistical Analysis 1: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p = 0.0007, Mixed Models Analysis; Least Squares Mean Difference = -1.1273, Standard Error of Mean 0.32552

5. Primary Outcome: Change From Baseline in Key Skin Biomarker Interleukin (IL)-13 Expression in Target Lesions Treated With Crisaborole Ointment 2% or Vehicle at Day 15
Description: IL-13 is one of the key skin biomarkers of atopic dermatitis. Expression levels tested by TLDA RT PCR were normalized to the housekeeping gene RPLP0 and log2-transformed prior to analysis.
Time Frame: Baseline (Day 1), Day 15
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log2(normalized expression)
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
log2(normalized expression) | -0.5484 (0.25767) | 0.2128 (0.27893)
Statistical Analysis 1: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p = 0.0871, Mixed Models Analysis; Least Squares Mean Difference = -0.7612, Standard Error of Mean 0.44266

6. Primary Outcome: Change From Baseline in Key Skin Biomarker Keratin 16 (KRT16) Expression in Target Lesions Treated With Crisaborole Ointment 2% or Vehicle at Day 15
Description: KRT16 is one of the key skin biomarkers of atopic dermatitis. Expression levels tested by TLDA RT PCR were normalized to the housekeeping gene RPLP0 and log2-transformed prior to analysis.
Time Frame: Baseline (Day 1), Day 15
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log2(normalized expression)
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
log2(normalized expression) | -2.4495 (0.30229) | -1.0854 (0.33131)
Statistical Analysis 1: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p = 0.0055, Mixed Models Analysis; Least Squares Mean Difference = -1.3641, Standard Error of Mean 0.48603

7. Primary Outcome: Change From Baseline in Key Skin Biomarker Elafin/Peptidase Inhibitor 3 (PI3) Expression in Target Lesions Treated With Crisaborole Ointment 2% or Vehicle at Day 15
Description: Elafin/PI3 is one of the key skin biomarkers of atopic dermatitis. Expression levels tested by TLDA RT PCR were normalized to the housekeeping gene RPLP0 and log2-transformed prior to analysis.
Time Frame: Baseline (Day 1), Day 15
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log2(normalized expression)
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
log2(normalized expression) | -2.4235 (0.33463) | -1.2989 (0.35218)
Statistical Analysis 1: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p = 0.0238, Mixed Models Analysis; Least Squares Mean Difference = -1.1246, Standard Error of Mean 0.49359

8. Primary Outcome: Change From Baseline in Key Skin Biomarker S100 Calcium Binding Protein A12 (S100A12) Expression in Target Lesions Treated With Crisaborole Ointment 2% or Vehicle at Day 15
Description: S100A12 is one of the key skin biomarkers of atopic dermatitis. Expression levels tested by TLDA RT PCR were normalized to the housekeeping gene RPLP0 and log2-transformed prior to analysis.
Time Frame: Baseline (Day 1), Day 15
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log2(normalized expression)
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
log2(normalized expression) | -3.2762 (0.39686) | -1.2849 (0.40613)
Statistical Analysis 1: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p = 0.0042, Mixed Models Analysis; Least Squares Mean Difference = -1.9913, Standard Error of Mean 0.68659

9. Secondary Outcome: Change From Baseline in Expression of Other Skin Biomarker (Epidermal Thickness) in Target Lesions Treated With Crisaborole Ointment 2% or Vehicle at Day 15
Description: Epidermal thickness was one of the other skin biomarkers of atopic dermatitis and was studied using immunohistochemistry (IHC). Expression data were log2-transformed.
Time Frame: Baseline (Day 1), Day 15
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log2-scale micrometers
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
log2-scale micrometers | -0.2737 (0.10653) | -0.1779 (0.08229)

10. Secondary Outcome: Change From Baseline in Expression of Other Skin Biomarkers (CD11c, CD3, FceR1, Ki67, Langerin) in Target Lesions Treated With Crisaborole Ointment 2% or Vehicle at Day 15
Description: CD11c+ dendritic cells (DCs), CD3+ T cells, FcEpsilon + DCs, Ki 67+ cells, and langerin+ cells (for langerhans cells) were studied using IHC. These parameters were referred to as CD11c, CD3, FceR1, Ki67, langerin, respectively, in the outcome measure title above and data table below. Expression data were log2-transformed.
Time Frame: Baseline (Day 1), Day 15
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log2-scale cells per square millimeter
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
log2-scale cells per square millimeter
  CD11c | -0.4736 (0.18946) | -0.1694 (0.11081)
  CD3 | -0.6219 (0.15152) | -0.2642 (0.13959)
  FceR1 | -0.4226 (0.16068) | -0.1314 (0.16513)
  Ki67 | -1.0983 (0.21512) | -0.8971 (0.19918)
  Langerin | 0.3694 (0.27896) | 0.2779 (0.19645)

11. Secondary Outcome: Change From Baseline in Expression of Other Skin Biomarkers (CCL13, Etc) in Target Lesions Treated With Crisaborole Ointment 2% or Vehicle at Day 15
Description: TLDA RT PCR was used to analyze the following other skin biomarkers: CCL13, CCL20, CCL26, CRLF2, CXCL1, CXCL2, CXCL9, CXCL10, DEFB4A, filaggrin (FLG), FOXP3, IFNG, IL-1B, IL-2, IL-2RA, IL-5, IL-6, IL-8, IL-9, IL-10, IL-12A, IL-15, IL-15RA, IL-17A, IL-17F, IL-19, IL-22, IL-23A, IL-31, IL-32, LOR, MMP-12, PDE4A, PDE4B, PDE4D, PPL, RNA18SP5, S100A7, S100A8, and S100A9. Expression levels were normalized to the housekeeping gene RPLP0 and log2-transformed prior to analysis.
Time Frame: Baseline (Day 1), Day 15
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log2(normalized expression)
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
log2(normalized expression)
  CCL13 | -0.3095 (0.21520) | 0.0604 (0.20967)
  CCL20 | -0.2016 (0.23629) | 0.1088 (0.23212)
  CCL26 | 0.0231 (0.18602) | 0.1195 (0.22820)
  CRLF2 | -0.8058 (0.13728) | -0.2023 (0.14431)
  CXCL1 | -1.4174 (0.23956) | 0.1924 (0.32423)
  CXCL10 | -1.0779 (0.36531) | 0.6697 (0.37822)
  CXCL2 | -0.5462 (0.21129) | 0.1945 (0.20700)
  CXCL9 | -0.9941 (0.33692) | 0.7562 (0.39811)
  DEFB4A | -3.5331 (0.42635) | -1.3456 (0.46988)
  FLG | -0.2155 (0.18503) | -0.3670 (0.22285)
  FOXP3 | -0.5115 (0.12709) | -0.0273 (0.16057)
  IFNG | -0.5588 (0.34472) | 0.5737 (0.31138)
  IL-10 | -0.3773 (0.19458) | 0.2950 (0.17314)
  IL-15 | -0.2307 (0.12331) | 0.2193 (0.11761)
  IL-15RA | -0.0780 (0.10814) | 0.2110 (0.10624)
  IL-17A | -1.1577 (0.57223) | 0.7516 (0.59970)
  IL-17F | -1.9482 (0.79294) | 0.5309 (0.88038)
  IL-19 | -3.1946 (0.78012) | -0.8108 (0.75460)
  IL-1B | -0.5792 (0.21864) | 0.2808 (0.29124)
  IL-2 | -0.5352 (0.26229) | 0.2769 (0.16896)
  IL-22 | -1.4970 (0.39951) | -0.0170 (0.35503)
  IL-2RA | -0.8836 (0.19462) | -0.0824 (0.22176)
  IL-31 | -1.5885 (0.60512) | -0.3997 (0.65363)
  IL-32 | -0.2992 (0.16762) | 0.1878 (0.15632)
  IL-5 | -0.3487 (0.51329) | -0.4148 (0.42311)
  IL-6 | -0.8814 (0.32670) | 0.1724 (0.36369)
  IL-8 | -1.9805 (0.37922) | -0.1698 (0.42603)
  IL-9 | -2.2803 (0.71683) | -1.0530 (0.68305)
  IL-12A | 0.2787 (0.20557) | 0.5251 (0.16751)
  IL-23A | -1.2754 (0.26058) | -0.1173 (0.28133)
  LOR | 0.3759 (0.19707) | -0.1041 (0.21965)
  MMP-12 | -1.9588 (0.39817) | -0.4205 (0.34033)
  PDE4A | 0.0105 (0.12015) | 0.1359 (0.11153)
  PDE4B | -0.1900 (0.12061) | 0.1923 (0.10897)
  PDE4D | -0.3865 (0.12920) | 0.0736 (0.12231)
  PPL | -0.3000 (0.09781) | -0.1933 (0.12180)
  RNA18SP5 | 0.1121 (0.08576) | -0.0221 (0.06550)
  S100A7 | -2.1764 (0.30729) | -0.8782 (0.26498)
  S100A8 | -2.4454 (0.36057) | -1.0669 (0.33255)
  S100A9 | -2.6155 (0.35209) | -1.2976 (0.33324)

12. Secondary Outcome: Number of Participants With Categorical Filaggrin (FLG) Expression at Day 15
Description: FLG expression was studied using IHC and categorized as no change, partial normalization, full normalization, or worsening by a blinded expert pathologist based on visual scoring.
Time Frame: Day 15
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
Participants
  No change | 10 | 19
  Partial normalization | 10 | 5
  Full normalization | 12 | 4
  Worsening | 7 | 11

13. Secondary Outcome: Number of Participants With Categorical Histological Response at Day 15
Description: Histological response was studied using IHC and categorized as non-responder or responder by a blinded expert pathologist based on a global assessment of all thickness, KRT16 and FLG stains.
Time Frame: Day 15
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
Participants
  Non-responder | 18 | 30
  Responder | 21 | 9

14. Secondary Outcome: Number of Participants With Categorical KRT16 Expression at Day 15
Description: KRT16 expression was studied using IHC and categorized as no change, slight improvement, good improvement, excellent improvement, or worsening by a blinded expert pathologist based on visual scoring.
Time Frame: Day 15
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 39 | 39
Participants
  No change | 13 | 18
  Slight improvement | 3 | 10
  Good improvement | 8 | 5
  Excellent improvement | 12 | 1
  Worsening | 3 | 5

15. Secondary Outcome: Change From Baseline in Lesion Severity as Measured by TSS at Day 8
Description: as for outcome 1
Time Frame: Baseline (Day 1), Day 8
Population: All randomized participants who received at least 1 dose of investigational product.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 40 | 40
units on a scale | -3.3 (0.36) | -1.2 (0.27)
Statistical Analysis 1: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -2.1, 95% CI 2-sided [-2.7 to -1.4], Standard Error of Mean 0.33

16. Secondary Outcome: Change From Baseline in Lesion Severity as Measured by Investigator Static Global Assessment (ISGA) at Day 8 and Day 15
Description: The lesion ISGA is an assessment of target lesion severity of atopic dermatitis. The lesion ISGA score ranges from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe), with higher score representing greater severity.
Time Frame: Baseline (Day 1), Days 8 and 15
Population: "Number of Participants Analyzed" signifies the number of participants who received at least 1 dose of investigational product. "Number Analyzed" refers to the number of evaluable participants for specified time points.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 40 | 40
units on a scale
  Day 8 | -1.3 (0.16) | -0.4 (0.11)
  Day 15: number analyzed (Participants) | 39 | 39
  Day 15 | -1.9 (0.15) | -0.8 (0.16)
Statistical Analysis 1: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Square Mean Difference = -0.9, 95% CI 2-sided [-1.3 to -0.6], Standard Error of Mean 0.17 — Comparison at Day 8
Statistical Analysis 2: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = -1.1, 95% CI 2-sided [-1.4 to -0.8], Standard Error of Mean 0.16 — Comparison at Day 15

17. Secondary Outcome: Change From Baseline in Lesion Severity as Measured by Pruritus Numerical Rating Scale (NRS) at Each Visit up to Day 15
Description: The intensity of pruritus was assessed by an NRS, which was a numeric rating scale ranging from 0 (no itching) to 10 (worst imaginable itching), with higher score indicating greater severity.
Time Frame: Baseline (Day 1), Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, and 15
Population: as for outcome 16
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 40 | 40
units on a scale
  Day 2: number analyzed (Participants) | 39 | 39
  Day 2 | -1.9 (0.36) | -1.0 (0.31)
  Day 3: number analyzed (Participants) | 39 | 39
  Day 3 | -2.2 (0.36) | -0.9 (0.38)
  Day 4 | -2.4 (0.33) | -1.1 (0.33)
  Day 5: number analyzed (Participants) | 38 | 38
  Day 5 | -2.7 (0.31) | -1.1 (0.36)
  Day 6: number analyzed (Participants) | 39 | 39
  Day 6 | -2.6 (0.34) | -1.3 (0.36)
  Day 7: number analyzed (Participants) | 39 | 39
  Day 7 | -3.1 (0.36) | -1.5 (0.35)
  Day 8: number analyzed (Participants) | 39 | 39
  Day 8 | -3.4 (0.35) | -1.5 (0.33)
  Day 9: number analyzed (Participants) | 39 | 39
  Day 9 | -3.4 (0.32) | -1.5 (0.34)
  Day 10: number analyzed (Participants) | 39 | 39
  Day 10 | -3.5 (0.34) | -1.6 (0.32)
  Day 11: number analyzed (Participants) | 37 | 37
  Day 11 | -3.5 (0.41) | -2.0 (0.41)
  Day 12: number analyzed (Participants) | 39 | 39
  Day 12 | -3.7 (0.40) | -1.5 (0.36)
  Day 13: number analyzed (Participants) | 39 | 39
  Day 13 | -4.0 (0.38) | -2.2 (0.39)
  Day 14: number analyzed (Participants) | 39 | 39
  Day 14 | -3.9 (0.36) | -2.2 (0.37)
  Day 15: number analyzed (Participants) | 39 | 39
  Day 15 | -3.9 (0.38) | -2.0 (0.41)
Statistical Analysis 1: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p = 0.0188, Mixed Models Analysis; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-1.6 to -0.1], Standard Error of Mean 0.36 — Comparison at Day 2
Statistical Analysis 2: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p = 0.0014, Mixed Models Analysis; Least-Square Mean of Difference = -1.2, 95% CI 2-sided [-1.9 to -0.4], Standard Error of Mean 0.36 — Comparison at Day 3
Statistical Analysis 3: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Least-Square Mean of Difference = -1.3, 95% CI 2-sided [-2.0 to -0.6], Standard Error of Mean 0.36 — Comparison at Day 4
Statistical Analysis 4: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square Mean of Difference = -1.5, 95% CI 2-sided [-2.2 to -0.8], Standard Error of Mean 0.36 — Comparison at Day 5
Statistical Analysis 5: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Least-Square Mean of Difference = -1.3, 95% CI 2-sided [-2.0 to -0.6], Standard Error of Mean 0.36 — Comparison at Day 6
Statistical Analysis 6: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square Mean of Difference = -1.5, 95% CI 2-sided [-2.3 to -0.8], Standard Error of Mean 0.36 — Comparison at Day 7
Statistical Analysis 7: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square Mean of Difference = -1.8, 95% CI 2-sided [-2.5 to -1.1], Standard Error of Mean 0.36 — Comparison at Day 8
Statistical Analysis 8: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square Mean of Difference = -1.9, 95% CI 2-sided [-2.6 to -1.2], Standard Error of Mean 0.36 — Comparison at Day 9
Statistical Analysis 9: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square Mean of Difference = -2.0, 95% CI 2-sided [-2.7 to -1.3], Standard Error of Mean 0.36 — Comparison at Day 10
Statistical Analysis 10: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square Mean of Difference = -1.6, 95% CI 2-sided [-2.3 to -0.9], Standard Error of Mean 0.37 — Comparison at Day 11
Statistical Analysis 11: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square Mean of Difference = -2.2, 95% CI 2-sided [-2.9 to -1.5], Standard Error of Mean 0.36 — Comparison at Day 12
Statistical Analysis 12: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square Mean of Difference = -1.9, 95% CI 2-sided [-2.6 to -1.2], Standard Error of Mean 0.36 — Comparison at Day 13
Statistical Analysis 13: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square Mean of Difference = -1.7, 95% CI 2-sided [-2.4 to -1.0], Standard Error of Mean 0.36 — Comparison at Day 14
Statistical Analysis 14: Comparison: Crisaborole Ointment 2% Treated Lesion vs Vehicle Treated Lesion; Crisaborole ointment 2% was superior to vehicle if p-value was <0.05; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square Mean of Difference = -1.9, 95% CI 2-sided [-2.7 to -1.2], Standard Error of Mean 0.36 — Comparison at Day 15

18. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) by Treatment Groups
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. AEs included both SAEs and non-serious AEs. Treatment-emergent AEs were those with initial onset or increasing in severity on or after the first dose of study treatment. Each participant received both crisaborole (for one target lesion) and vehicle (for the other target lesion) on the same days during double-blind period, and only crisaborole during open-label period; therefore AEs were reported for each treatment group for participants to capture all AEs, instead of each treatment for treated area as it only captures AEs occurred at treated areas (see next Outcome Measure).
Time Frame: From first dose of study treatment up to Day 71
Population: All participants in each treatment group who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Crisaborole Ointment 2% + Vehicle in Double-Blind Period: On Days 1 to 14, for each participant, one target lesion was treated with crisaborole ointment 2% and the other target lesion was treated with vehicle, i.e., each participant was treated with both crisaborole and vehicle. This reporting group represents the participants who were treated with both crisaborole ointment 2% and vehicle during Days 1 to 14.
- Crisaborole Ointment 2% in Open-Label Period: On Days 15 to 42, each participant received crisaborole ointment 2% for all atopic dermatitis skin areas (excluding scalp).
Arm/Group | Crisaborole Ointment 2% + Vehicle in Double-Blind Period | Crisaborole Ointment 2% in Open-Label Period
Number analyzed (Participants) | 40 | 39
Participants
  Treatment-emergent AEs | 27 | 16
  Treatment-emergent SAEs | 0 | 0

19. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) by Medical Dictionary for Regulatory Activities (MedDRA) Preferred Term, Which Occurred in the Treatment Area During the Double-Blind Period
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Treatment-emergent AEs were those with initial onset or increasing in severity on or after the first dose of study treatment. During double-blind period, there were a total of 2 treatment areas (for target lesions) for each participant. For this outcome measure, treatment-emergent AEs occurred at each treated area during double-blind period were summarized. MedDRA version 21.0 coding dictionary was used.
Time Frame: From first dose of study treatment (on Day 1) to Day 15 skin biopsy collection
Population: This outcome measure was summarized by the treatment areas during the double-blind period; therefore, the analysis population here represents the participants who received at least 1 dose of investigational product for each treatment area in double-blind period.
Measure: Count of Participants; unit: Participants
Arm/Group | Crisaborole Ointment 2% Treated Lesion | Vehicle Treated Lesion
Number analyzed (Participants) | 40 | 40
Participants
  Application site dermatitis | 0 | 1
  Application site erythema | 1 | 0
  Application site pain | 2 | 4
  Application site pruritus | 1 | 2
  Application site folliculitis | 1 | 0
  Post procedural haemorrhage | 0 | 1
  Procedural pain | 2 | 2
  Suture related complication | 1 | 2

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to Day 71
Description: Each participant received both crisaborole (for one target lesion) and vehicle (for the other target lesion) on the same days during double-blind period, and only crisaborole during open-label period; therefore AEs were reported for each treatment group for participants to capture all AEs, instead of each treatment for treated area as it only captures AEs occurred at treated areas (see Outcome Measure 19 for the treated area AEs).
Arm/Group | Crisaborole Ointment 2% + Vehicle in Double-Blind Period | Crisaborole Ointment 2% in Open-Label Period
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 27/40 | 16/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crisaborole Ointment 2% + Vehicle in Double-Blind Period (N=40) | Crisaborole Ointment 2% in Open-Label Period (N=39)
Application site pain (General disorders) | 4 | 4
Gastroenteritis (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 7 | 5
Procedural pain (Injury, poisoning and procedural complications) | 6 | 1
Suture related complication (Injury, poisoning and procedural complications) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 8 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 5
Noninfective conjunctivitis (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Application site dermatitis (General disorders) | 1 | 0
Application site erythema (General disorders) | 1 | 0
Application site paraesthesia (General disorders) | 0 | 1
Application site pruritus (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Application site folliculitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Graft complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT03233529/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03233529/SAP_001.pdf